CLINICAL TRIAL: NCT06446856
Title: EVEN - Effects of VR on Empathy for Nature in Patients with Psychosis and Depressive Disorders / Effekte Von Virtueller Realität (VR) Auf Naturverbundenheit Und Empathie in Patient:innen Mit Psychotischen Und Depressiven Erkrankungen
Brief Title: EVEN - Effects of VR on Empathy for Nature in Patients with Psychosis and Depressive Disorders
Acronym: EVEN
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Universität Potsdam, Department Erziehungswissenschaft, Arbeitsbereich Schulbezogene Medienbildung (Unknown)
Responsible Party: Principal Investigator, Alva Lütt, Dr. med. Alva Lütt, MD, Charite University, Berlin, Germany
Other Study IDs: EA2/046/24
Record Dates: First submitted 2024-05-25; First posted 2024-06-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Depressive Disorder; Schizophrenia; Healthy Control
MeSH Terms: conditions — Depressive Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- VR study group: 20 patients with depressive disorder
  Interventions: Device: VR application
- VR active control group: 20 patients with psychotic disorder.
  Interventions: Device: VR application
- VR healthy control group: 20 patients with no psychiatric disorder
  Interventions: Device: VR application

INTERVENTIONS:
Device: VR application — The VR application consists of a software ("Tree") developed as part of a research project at MIT and legally acquired via the HTC store Viveport. Duration of the VR application: approx. 5 min.

SUMMARY:
Study group: Experimental study to evaluate empathy, compassion, and nature connectedness before and after an immersive virtual reality experience in patients with depressive disorder, patients with psychotic disorder and healthy control subjects (subjects between 18 and 65 years of age).

Primary hypothesis: The increase in nature connectedness explored by virtual body ownership of a tree in VR differs depending on the health condition (schizophrenia, depression, healthy controls).

ELIGIBILITY:
Inclusion Criteria:

* age: 18-65 years
* Inpatients and outpatients treated at the Psychiatric University Clinic of the Charité at St.

Hedwig Hospital

* diagnosis of depressive disorder (ICD-10: F32.X, F33.X) or diagnosis of schizophrenia (F20.X) or healthy controls without psychiatric diagnosis
* able to provide written informed consent

Exclusion Criteria:

* Acute suicidality or danger to others
* Primarily treatment-requiring eating disorder
* Acute dermatological condition affecting the hands that can distort skin conductivity measurements
* Control group: psychiatric or psychosomatic pre-diagnoses (except for the psychiatric active control group), other exclusion diagnoses corresponding to the patient group

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with depressive or psychotic disorder treated in the inpatient or outpatient psychiatric clinics or day clinics of the Psychiatric University Hospital Charité at St. Hedwig-Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Nature Connectedness | For all groups pre and directly post VR exposure
  Measurement of Nature Connectedness as a state with the "Inclusion of Nature in Self" (INS)-Questionnaire (Kleespies et al., 2021), pre and post VR exposure.

SECONDARY OUTCOMES:
Empathy | For all groups pre and directly post VR exposure (within the same session of 1 hour)
  Evaluation of empathy with the Multifaceted Empathy Test (MET; (Dziobek et al., 2008) pre and post VR exposure
Compassion | For all groups pre and directly post VR exposure (within the same session of 1 hour)
  Evaluation of Compassion (state compassion) pre and post VR exposure with the Positive and Negative Affect Schedule (PANAS) and five integrated items measuring compassion based on Pfattheicher et al., 2015.
symptom burden | For the VR study group (patients with depressive disorder) and VR active control group (patients with psychotic disorder) pre and post VR exposure (within the same session of 1 hour)
  Measured with the PANAS (see above) and with the Visual Analogue Scale (0-10) measuring the burden of the 3 main symptoms, previously specified during assessment of symptom severity (PANSS; (Kay et al., 1987) and Beck Depression Inventory (BDI, Beck et al., 1961))
Embodiment - Feeling of virtual body ownership | post VR exposure for all groups (within the same session of 1 hour)
  Evaluation with a subscale of the Embodiment scale by Ahn et al. (2016) adapted from Slater et al. (2010)
Spirituality | pre VR exposure for all groups
  Evaluation of spirituality using the 4-item short version of the questionnaire "Transpersonales Vertrauen" (Hampel et al., 2019) pre VR exposure.
Presence in VR | post VR exposure for all groups (within the same session of 1 hour)
  Scale according to Ahn et al. (Ahn et al., 2016), adapted from the "Spatial Presence scale" by Bailenson et al. (2005) - own German translation adapted to the virtual Amazon forest area (Spangenberger et al., 2024)
Virtual Reality Simulator Sickness | post VR exposure for all groups (within the same session of 1 hour)
  Cyber Sickness as a potential side effect of VR, measured with the Virtual Reality Sickness Questionnaire (Kim et al., 2018)
Explorative evaluation of electrodermal activity (EDA) | during (approx. 5 minutes) VR exposure
  Explorative evaluation of electrodermal activity (EDA), e.g., skin conductance level (SCL) and skin conductance responses (SCR) in micro siemens during VR exposure

OTHER OUTCOMES:
demographic variables | pre VR exposure for all groups
  acquisition of demographic data
comorbidities | pre VR exposure for all groups
  acquisition of psychiatric comorbidities and physical illnesses
symptom severity - psychotic symptoms | For the VR study group (patients with depressive disorder) and VR active control group (patients with psychotic disorder) pre VR exposure (within the same session of 1 hour)
  Assessment of symptom severity with the Positive and Negative Syndrome Scale (PANSS; Kay et al., 1987)
symptom severity - depressive symptoms | For the VR study group (patients with depressive disorder) and VR active control group (patients with psychotic disorder) pre VR exposure (within the same session of 1 hour)
  Assessment of symptom severity with the Beck Depression Inventory (BDI; Beck et al., 1961)

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital Charité at St. Hedwig Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided